CLINICAL TRIAL: NCT07195994
Title: A Randomized, Single-blind, Controlled, Parallel Clinical Trial to Examine the Efficacy and Safety of an Investigational Product With and Without Use of Semaglutide on Glycemic Response in Adults With Prediabetes or Type 2 Diabetes
Brief Title: A Clinical Trial to Examine the Efficacy and Safety of an Investigational Product With and Without Use of Semaglutide on Glycemic Response in Adults With Prediabetes or Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: QuickSilver Scientific (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24QSCFA02
Record Dates: First submitted 2025-09-18; First posted 2025-09-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-06

CONDITIONS: Prediabetes / Type 2 Diabetes
Keywords: Prediabetes; AMPK Charge+®; Semaglutide; GLP-1 agonist
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind clinical trial wherein the Statistician and Research Scientist will be blinded to the allocation of study arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMPK Charge+® (Experimental): AMPK Charge+® is a dietary supplement comprised of highly purified phospholipids, diindolylmethane, quercetin dihydrate, milk thistle seed extract, resveratrol, and berberine delivered using liposomal and nanoemulsion technology.
  Interventions: Dietary Supplement: AMPK Charge+®
- AMPK Charge+® with semaglutide (Active Comparator): Subcutaneous semaglutide (Ozempic®), a glucagon-like peptide-1 (GLP-1) receptor agonist, is indicated for adults with T2D to improve glycemic control with the safety and efficacy extensively investigated leading to approvals by the United States (U.S.) Food and Drug Administration and Health Canada
  Interventions: Dietary Supplement: AMPK Charge+® with semaglutide

INTERVENTIONS:
Dietary Supplement: AMPK Charge+® — Participants will be instructed to consume 1 teaspoon (5 mL) on an empty stomach before breakfast and 1 teaspoon on an empty stomach in the afternoon and to hold the product in the mouth for approximately 30-90 seconds before swallowing starting on Day 1.
  Arms: AMPK Charge+®
Dietary Supplement: AMPK Charge+® with semaglutide — Participants will be instructed to use the provided measuring tool to take 1 teaspoon (5 mL) on an empty stomach before breakfast and 1 teaspoon on an empty stomach in the afternoon and to hold the product in the mouth for approximately 30-90 seconds before swallowing starting on Day 1. Participants will be instructed to administer subcutaneous semaglutide once per week beginning with a dose of 0.25 mg for four weeks at which point participants will be instructed to increase the dose to 0.5 mg per week for the remainder of the study period.
  Arms: AMPK Charge+® with semaglutide

SUMMARY:
This is a randomized, single-blind, controlled, parallel clinical trial to examine the efficacy and safety of AMPK Charge+® with and without use of semaglutide on glycemic response in adults with prediabetes or Type 2 Diabetes. The main question it aims to answer is:

What is the difference in change in fasting blood glucose and insulin, and hemoglobin A1c (HbA1c) from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide?

Participants will consume AMPK Charge+® with or without semaglutide injections and will be evaluated for glycemic response parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Males & females between 18 years of age or older
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if becomes sexually active during this study
3. Individuals eligible for, but not currently taking, semaglutide therapy as per standard-of-care including adults with:

   1. Prediabetes (HbA1c 6.0-6.5%) who are treatment naïve
   2. Type 2 Diabetes (HbA1c 6.5-7.5%) who are treatment naïve and metformin is inappropriate due to contraindication or intolerance
4. Self-reported stable body weight defined as not having gained or lost more than 5 kg of body weight in the three months prior to baseline
5. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, sleep, use of nicotine, tobacco and cannabinoid products) as much as possible throughout the study
6. Willingness to complete questionnaires, records, and diaries associated with the study and to complete all clinic visits
7. Provided voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, intolerance, or dietary restriction preventing use of study products
3. Personal or family history of MTC or in patients with MEN 2
4. Unstable metabolic disease or chronic diseases as assessed by the QI
5. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
6. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI (See Section 7.3)
7. Type I diabetes or diabetic ketoacidosis
8. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
9. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
10. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
11. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
12. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
13. Individuals with an autoimmune disease or are immune compromised
14. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
15. Self-reported confirmation of blood/bleeding disorders as assessed by the QI
16. Alcohol intake average of >2 standard drinks per day as assessed by the QI
17. Alcohol or drug abuse within the last 12 months
18. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy and/or safety of the study products (See Section 7.3)
19. Clinically significant abnormal laboratory results at screening as assessed by the QI
20. Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
21. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
22. Individuals who are unable to give informed consent
23. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The difference in change in fasting blood glucose between AMPK Charge+® and AMPK Charge+® with semaglutide | Day 0 to 84
  The difference in change in fasting blood glucose from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide
The difference in change in fasting insulin between AMPK Charge+® and AMPK Charge+® with semaglutide | Day 0 to 84
  The difference in change in fasting insulin from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide
The difference in change in hemoglobin A1c (HbA1c) between AMPK Charge+® and AMPK Charge+® with semaglutide | Day 0 to 84
  The difference in change in hemoglobin A1c (HbA1c) from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide

SECONDARY OUTCOMES:
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in fasting blood glucose | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in fasting blood glucose
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in HbA1c | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in fasting HbA1c
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in fasting insulin | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in fasting insulin
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in Total Cholesterol (TC),
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in Total Cholesterol (TC),
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR) | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in Low-Density Lipoprotein (LDL) cholesterol
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in High-Density Lipoprotein (HDL) cholesterol | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in High-Density Lipoprotein (HDL) cholesterol
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in , High-Density Lipoprotein (HDL) cholesterol | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in , High-Density Lipoprotein (HDL) cholesterol
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Triglycerides (TG), | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in Triglycerides (TG),
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Triglycerides (TG), | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in ,Triglycerides (TG),
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in TC:HDL-C, TG:HDL-C, and LDL-C:HDL-C ratios | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in TC:HDL-C, TG:HDL-C, and LDL-C:HDL-C ratios
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in TC:HDL-C, TG:HDL-C, and LDL-C:HDL-C ratios | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in TC:HDL-C, TG:HDL-C, and LDL-C:HDL-C ratios
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Apolipoprotein B100 (ApoB100) | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in Apolipoprotein B100 (ApoB100)
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Inflammatory markers as assessed by C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR) | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in Inflammatory markers as assessed by C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR)
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in Inflammatory markers as assessed by C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR) | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in Inflammatory markers as assessed by C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR)
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in e. Body weight | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in e. Body weight
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in e. Body weight | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in e. Body weight
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in f. Framingham 10-year cardiovascular risk score (FCVRS) | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in f. Framingham 10-year cardiovascular risk score (FCVRS)
The difference in change between AMPK Charge+® and AMPK Charge+® with semaglutide in f. Framingham 10-year cardiovascular risk score (FCVRS) | Day 0 to 42
  The difference in change from baseline at Day 42 between AMPK Charge+® and AMPK Charge+® with semaglutide in f. Framingham 10-year cardiovascular risk score (FCVRS)
The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in Postprandial glucose and insulin as assessed by an oral glucose tolerance test (OGTT) | Day 0 to 84
  The difference in change from baseline at Day 84 between AMPK Charge+® and AMPK Charge+® with semaglutide in Postprandial glucose and insulin as assessed by an oral glucose tolerance test (OGTT)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada